CLINICAL TRIAL: NCT06591936
Title: Genetic Profile of Alpha Thalassemia Children at Sohag University Hospital .
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Abdelrahim, Resedent doctor , pediatric and neonatology, Sohag University
Other Study IDs: soh-med-24-08-02MS
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alpha-Thalassemia
MeSH Terms: conditions — alpha-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- genetic of alpha thalathemia

SUMMARY:
Genetic profile of alpha thalassemia children at sohag university hospital ,the aim to determine the prevelance , molecular character of the disorder, characterized by decreased synthesis of alpha -globin Recent work to provide mechanisms for phenotypic heterogeneity .

ELIGIBILITY:
Inclusion Criteria:

* Acase suspecteed of alpha thalassemia
* age between 0-18years
* micocytic hypochromic anemia not iron deficiency anemia or Beta thalassemia

Exclusion Criteria:

* Age more than 18 years
* healthy children free from any chronic hematological disease
* micocytic hypochromic anemia either iron deficiency anemia or Beta thalassemia

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Acase suspecteed of alpha thalassemia
  * age between 0-18years
  * micocytic hypochromic anemia not iron deficiency anemia or Beta thalassemia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
PCR for prevelance of mutation phenotype | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code
Time Frame: one year